CLINICAL TRIAL: NCT03545347
Title: Preliminary Effect and Safety of Physiotherapy With Strength Training and Protein-rich Nutritional Supplement in Combination With Anabolic Steroids in Cross-continuum Rehabilitation of Patients With Hip Fracture - a Randomized Controlled Pilot Trial. (The HIP-SAP Trial)
Brief Title: Physiotherapy, Nutritional Supplement and Anabolic Steroids in Rehabilitation of Patients With Hip Fracture.
Acronym: HIP-SAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morten Tange Kristensen PT, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Tange Kristensen PT, PhD, Senior Researcher, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HvidovreUH-HIP-SAP-1; 2017-001543-13 (EudraCT Number)
Record Dates: First submitted 2018-05-18; First posted 2018-06-04 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Hip Fractures
Keywords: Rehabilitation; Physiotherapy; Strength training; Anabolic steroids; Nutritional supplement
MeSH Terms: conditions — Hip Fractures | interventions — Nandrolone Decanoate; Nandrolone; Anabolic Androgenic Steroids; Physical Therapy Modalities; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nandrolone Decanoate (Experimental): Physical therapy with strength training, protein-rich nutritional supplement plus Nandrolone decanoate.
  Interventions: Drug: Nandrolone Decanoate; Dietary Supplement: Protein-rich nutritional supplement; Other: Physical therapy
- Placebo (Sodium Chloride) (Placebo Comparator): Physical therapy with strength training, protein-rich nutritional supplement plus placebo.
  Interventions: Dietary Supplement: Protein-rich nutritional supplement; Other: Physical therapy; Drug: Sodium Chloride 9mg/ml Injection

INTERVENTIONS:
Drug: Nandrolone Decanoate — Injections every 3 weeks, last injection at week 12. Women 50 mg, men with total testosterone ≥ 11 nmol/l will receive 100 mg, and men with total testosterone < 11 nmol/l will receive a dose of 200 mg.
  Other Names: Deca-durabolin; anabolic steroid
  Arms: Nandrolone Decanoate
Dietary Supplement: Protein-rich nutritional supplement — The protein-rich nutritional supplement is a liquid containing 18 g milk-based protein pr bottle. Patients will receive a minimum of 1.35 g/kg bodyweight/day); which means that most patients will receive 2 bottles per day for 12 weeks.
  Other Names: Nestle Resource fiber 2.0
Other: Physical therapy — The physical therapy intervention will include progressive strength training initiated daily on weekdays during hospitalization and continued twice per week in the outpatient rehabilitation program in the municipality (treatment as usual but with strength training as an obligatory component) for a total intervention period of 12 weeks from time of inclusion.
  Other Names: Physiotherapy
Drug: Sodium Chloride 9mg/ml Injection — Placebo injection of 1 ml Sodium Chloride
  Other Names: Saline
  Arms: Placebo (Sodium Chloride)

SUMMARY:
This pilot trial investigates the preliminary effect and safety of a 12 week multi-modal intervention initiated during admission in the acute ward after hip fracture surgery. The intervention under investigation is a combination therapy consisting of physiotherapy, protein-rich nutritional supplement and nandrolone decanoate (Deca-Durabolin) supplement. The investigators expect the combination therapy to be a preliminary effective and safe treatment in elderly patients with hip fracture and that this combination therapy intervention program is more efficacious in improving muscle strength, and physical function 14 weeks after hip fracture surgery, compared to physiotherapy, protein-rich nutritional supplement plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone surgery for a hip fracture at Amager-Hvidovre University Hospital and admitted at the Hip Fracture Unit at the hospital
* Age >=60 years
* Ability to speak and understand Danish and with a Danish Social Security Number
* Able to give written informed consent
* Residing at home and with an independent pre-fracture indoor walking ability (NMS≥2)

Exclusion Criteria:

* Postoperative weight-bearing restrictions
* Multiple fractures
* Active cancer or suspected pathological fracture
* Patients unable/unwilling to cooperate to testing and rehabilitation
* Planned/elective hospitalization within the trial period.
* Cognitive dysfunction determined by chart review, reported by nursing staff, or observed by trained research staff (disoriented, dementia, active delirium)
* Uncontrolled blood pressure (systolic > 150 mmHg, or diastolic > 100 mmHg)
* Heart disease in the form of peri-, myo- or endocarditis.
* History of stroke with motor disability.
* Heart failure (NYHA class III and IV)
* Evidence of kidney failure or renal impairment (estimated glomerular filtration rate < 30 mL/min/1.73 m2 or serum creatinine >200μmol/L)
* Abnormal liver function tests (alanine aminotransferase, γ-glutamyltransferase, bilirubin, or alkaline phosphatase >2 times the upper limit of normal) or history of hepatic tumor.
* Elevated hematocrit ≥ 50%
* History of breast or prostate cancer
* Abnormally elevated serum PSA assesed at the 3 week control corresponding to PSA < 4.0 µg/L (60-70 years), PSA < 5.0 µg/L (>70 years).
* Allergic to any ingredient in the Deca-Durabolin solution (Nandrolone, benzyl alcohol, arachis oil (peanut-oil) and allergy to peanuts or soya) or milk protein allergy (related to the nutritional drink).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Change in maximal isometric knee-extension strength (Nm/Kg) in the fractured limb. | Baseline and 14 weeks after inclusion
  Measured using a belt fixed handheld dynamometer.

SECONDARY OUTCOMES:
Maximal isometric knee-extension strength (Nm/Kg) in the fractured limb in % of the non-fractured limb | Baseline and 14 weeks after inclusion
  Measured using a belt fixed handheld dynamometer.
Maximal isometric knee-extension strength (Nm/Kg) in the non-fractured limb. | Baseline and 14 weeks after inclusion.
  Measured using a belt fixed handheld dynamometer.
Hand-grip strength in the dominant hand. | Baseline and 14 weeks after inclusion.
  Measured using a handheld dynamometer, expressed in kg.
Bone mineral density (BMD) | Baseline and 14 weeks after inclusion.
  Registration of total body, total hip, femoral neck, lumbar spine. Assessed by Dual-energy X-ray absorptiometry (DEXA), expressed in g/cm2. Further the T-score is registered. The DEXA is conducted in accordance with the department's standard procedures.
Lean body mass (LBM) | Baseline and 14 weeks after inclusion.
  Registration of total body, legs bilaterally, arms bilaterally. Assessed by DEXA and expressed in kg.
Fat mass | Baseline and 14 weeks after inclusion.
  Total body. Assessed by DEXA and expressed in kg.
Nutrition screening using the Mini Nutritional Assessment Short Form (MNA-SF). | Baseline (prefracture) and 14 weeks after inclusion.
  Total score from 0-14 points, high scores indicating better nutritional status
Gait speed will be assessed using the 10 meter walk test (10mWT) | Baseline and 14 weeks after inclusion.
  The results reported in meters walked per second (m/s).
Timed up and go test (TUG) | Baseline and 14 weeks after inclusion.
  Performed using a 4 wheeled rollator and measured in seconds. The patient has to rise from a chair, walk 3 meters, turnaround, walk back and sit down.
The de Mortons Mobility Index (DEMMI) | Baseline and 14 weeks after inclusion.
  Measures mobility and consists of 15 mobility items ranging from mobility in bed to dynamic balance. The test results in a total score from 0 to 100 with 100 representing the highest level of mobility.
Upright time | Measured from the time of the control week 12 and one week ahead.
  Assessed by using a body-worn accelerometer-based activity monitor (ActivePAL). The monitor will be attached to the thigh. The patient will wear the monitor for 7 days.
Functional level is assessed by the New Mobility Score (NMS). | Baseline (prefracture) and 3/6/9/12/14 weeks after inclusion.
  The patients are interviewed about walking ability indoor, outdoor and when shopping. the week prior to hospital admission. The total score range from 0 to 9. A Higher score indicating higher independence.
The EQ-5D-3L is used for assessing health related quality of life. | Baseline (prefracture) and 14 weeks after inclusion
  It is administered via interview.
Hip fracture related pain at rest and during outcome assessment | Baseline and 3/6/9/12/14 weeks after inclusion.
  It is evaluated by Verbal Ranking Scale (VRS). The patient expresses pain levels on a verbal scale from 0-4, higher score indicating higher pain levels.
Global Rating of Change Scale | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Assessment of patient perceived change in walking ability during the trial period.
The Short Falls Efficacy Scale-International (Short FES-I) | Baseline and 14 weeks after inclusion.
  Measures the patient's fear of falling (Score 7-28, higher scores indicating a higher fear of falling). It is administered as an interview.
Fatigue is assessed using the Short Form (36) Health Survey (SF36) vitality subscale. | Baseline (prefracture), and 3/6/9/12/14 weeks after inclusion.
  The scale consists of 4 items related to fatigue/energy. Score range from 0-100 points; high score defines a more favorable health state. Administered as an interview.
Depression is assessed using the Geriatric Depression Scale (GDS-15) | Baseline (prefracture) and 14 weeks after inclusion.
  Administered as an interview. Score range 0-15.
Re-admissions | 14 weeks after inclusion.
  Assessed through the medical journal/interviews.
Residential status (including home care) | Baseline (prefracture) and 14 weeks after inclusion.
  Change in residential status and home care (help provided in the patients home). Assessed through the medical journal/interviews.
Mortality | 14 weeks after inclusion.
  Assessed through the medical journal/Danish civil register.
Falls | Assessed through weekly telephone interviews and hospital visits at 3/6/9/12/14 weeks after inclusion.
  Number of falls. Assessed through interviews
Total testosterone (nmol/l) | Baseline and 14 weeks after inclusion.
  Blood test
Luteinizing hormone (LH), IU/l | Baseline and 14 weeks after inclusion.
  Blood test
Follicle-stimulating hormone (FSH) IU/l | Baseline and 14 weeks after inclusion.
  Blood test
Sex hormone binding globulin (SHBG), nmol/l | Baseline and 14 weeks after inclusion.
  Blood test
Lipid profile (Total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride) mmol/l. | Baseline and 14 weeks after inclusion.
  Blood test
C-reactive protein (CRP), mg/l. | Baseline and 14 weeks after inclusion.
  Blood test
Hematocrit (B-Erythrocyte, vol.fr.) | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Hemoglobin | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Creatinine | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Carbamide | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Sodium (Na+) | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Potassium (K+) | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Calcium | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Liver tests (Albumin, Alanine aminotransferase (ALAT), γ-glutamyltransferase, Bilirubin) | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
International Normalized Ratio (INR) | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Prostate Specific Antigen (PSA) | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Glucose | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, blood test
Blood pressure | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Safety parameter, assessed using a 'Blood pressure monitor' (mmHg).
Facial hirsutism | Baseline, and 3/6/9/12/14 weeks after inclusion.
  Change in facial hair assessed using the 2 face-related items of Ferriman-Galway Hirsutism Score.
Hoarseness | Assessed at baseline and through weekly telephone interviews and hospital visits at 3/6/9/12/14 weeks after inclusion.
  Change in voice, reported by patient or observed by interviewer (no specific score available for this evaluation).
Other adverse events | Assessed through weekly interviews and hospital visits at 3/6/9/12/14 weeks after inclusion.
  Assessed through interview, observation
Edema in non-fractured leg | Assessed at baseline and through weekly interviews and hospital visits at 3/6/9/12/14 weeks after inclusion.
  Change in edema assessed through interview

CONTACTS AND LOCATIONS:
Overall Officials: Morten T Kristensen, PT, PhD, Study Director — Department of Occupational and Physical Therapy and Department of Orthopedic Surgery, Amager-Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hulsbaek S, Bandholm T, Ban I, Foss NB, Jensen JB, Kehlet H, Kristensen MT. Feasibility and preliminary effect of anabolic steroids in addition to strength training and nutritional supplement in rehabilitation of patients with hip fracture: a randomized controlled pilot trial (HIP-SAP1 trial). BMC Geriatr. 2021 May 20;21(1):323. doi: 10.1186/s12877-021-02273-z. PMID 34016037
- [Derived] Hulsbaek S, Ban I, Aasvang TK, Jensen JB, Kehlet H, Foss NB, Bandholm T, Kristensen MT. Preliminary effect and feasibility of physiotherapy with strength training and protein-rich nutritional supplement in combination with anabolic steroids in cross-continuum rehabilitation of patients with hip fracture: protocol for a blinded randomized controlled pilot trial (HIP-SAP1 trial). Trials. 2019 Dec 23;20(1):763. doi: 10.1186/s13063-019-3845-y. PMID 31870451